CLINICAL TRIAL: NCT03951259
Title: A Randomised, Double-blind, Placebo-controlled, Phase 2 Study Evaluating the Safety and Efficacy of SM934 in Adult Subjects With Active Systemic Lupus Erythematosus
Brief Title: Safety and Efficacy of SM934 Compared to Placebo in Adult Subjects With Active Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Jiangsu ZuoYou Medicine Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM934
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — beta-aminoarteether maleate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SM934 10mg (Experimental): SM934 10mg（1 tablet）+Placebo（4 tablets）p.o. qd in combination with steroids
  Interventions: Drug: SM934
- SM934 30mg (Experimental): SM934 10mg（3 tablet）+ Placebo（2 tablets）p.o. qd in combination with steroids
  Interventions: Drug: SM934
- SM934 50mg (Experimental): SM934 10mg（5 tablet）p.o. qd in combination with steroids
  Interventions: Drug: SM934
- Placebo (Placebo Comparator): Placebo（5 tablets）p.o. qd in combination with steroids
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: SM934 — In this study, the investigating intervention is oral administration of SM934. SM934 is a water-soluble derivative of arteminisin, which exerts immunosuppressive functions in vitro and in vivo.
  Arms: SM934 10mg; SM934 30mg; SM934 50mg
Drug: Placebos — The placebo pills are made identical to the investigating SM934 in appearance.
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, phase 2 study. The purpose of the study is to initially evaluate the safety and efficacy of SM934 combined with steroids compared to placebo in adult subjects with active systemic lupus erythematosus (SLE) over a 12-week period.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 70;
* Have a clinical diagnosis of SLE according to SLICC-2012 classification criteria;
* Have active SLE with SLEDAI-2k ≥ 6;
* Have positive anti-nuclear antibody (ANA) test results;
* Are on a stable steroids treatment (equals to prednison more than 7.5mg daily but no more than 0.5mg/kg/d) for SLE for at least 30 days prior to first dose of study agent;
* Females of childbearing age are willing to use appropriate contraception;
* Are voluntary to to provide and sign voluntary informed consent is given;

Exclusion Criteria:

* Have any unstable or progressive manifestation of SLE, including but not limited to Central nervous system (CNS) involvement, transverse myelitis, systemic vasculitis, vasculitis with GI involvement, severe or rapidly progressive lupus nephritis, lupus nephritis with proteinuria > 3g/24h, pulmonary hemorrhage, myocarditis;
* Have abnormal liver function test or renal function test: Alanine aminotransferase（ALT）or aspartate aminotransferase (AST) >2 upper limit of normal (ULN); Gamma-glutamyl transferase (GGT) >1.5 ULN; Creatinine or Blood urea nitrogen (BUN) >1.5 ULN;
* Have a history of acute myocardiac infarction, unstable angina, severe arrhythmias within 6 months prior to first dose of study agent;
* Have any major illness/condition or evidence of an unstable clinical condition not due to SLE (eg, cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, psychiatric), which, in the Investigator's judgment, will substantially increase the risk to the participant if he or she participates in the study;
* Have any acute or chronic infectious disease, which requires medical intervention;
* Have a history of cancer within the last 5 years, except for adequately treated skin cancer, or carcinoma in situ of the uterine cervix;
* Have a planned surgical procedure;
* Have received a biologic investigational agent in the past one year;
* Have received the following treatment within 30 days prior to first dose of study agent: live vaccine; change of glucocorticoids dose; IV, intra-muscular (IM), intra-articular (IA) administration of glucocorticoids; other immunosuppressants/immunomodulators; anti-malarial drugs; traditional medicines which has proved to be effective in SLE;
* Have had a major organ transplant;
* Have a history of HIV, or test positive at screening for HIV;
* Test positive for Hepatitis B virus (HBV)-DNA or Hepatitis C virus (HCV)-RNA;
* Have or have had a substance abuse (drug, alcohol) problem in the past one year;
* Are currently using or planned to use estrogen-containing contraceptive methods;
* Have enrolled in an investigational study within 3 months prior to first dose of study agent;
* Investigator considers candidates not appropriating for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Percentage of Subjects with Lupus Low Disease Activity Score (LLDAS) in each group | Week 12
  LLDAS is defined as meeting the following criteria:
  1. SLEDAI-2K ≤4, with no activity in major organ systems (renal, CNS, cardiopulmonary, vasculitis), and no reported fever, hemolytic anemia, or gastrointestinal activity)
  2. No new disease activity compared with the previous assessment (no new British isles lupus assessment group (BILAG) A domain score or no more than 1 new BILAG B domain score)
  3. PGA ≤1 on a 0-3 scale visual visual analogue scale (VAS)
  4. A current prednisone (or equivalent) dose of ≤7.5 mg daily
  5. Well-tolerated standard maintenance doses of permitted immunosuppressive drugs
Percentage of Subjects with Systemic Lupus Erythematosus Responder Index - 4 (SRI-4) response in each group | Week 12
  SRI-4 response is defined as:
  1. ≥ 4-point reduction from baseline in SLEDAI-2K score
  2. No new BILAG A and no more than 1 new BILAG B domain score
  3. No worsening from baseline in the PGA (<10% worsening from baseline).
Percentage of Subjects with Treatment-Emergent Adverse Events (TEAEs) in each group | Baseline through Week 13
  Percentage of Subjects with TEAEs in each group

SECONDARY OUTCOMES:
Percentage change of SLEDAI-2000 and Physician Global Assessment (PGA) from baseline in each group | Week 12
  Percentage change of SLEDAI-2000 and PGA from baseline in each group
Percentage of Subjects with 30% improvement in Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) score in each group | Week 12
  Percentage of subjects who have at least 30% improvement in CLASI score compared to baseline.
Change of SLICC/ACR from baseline | Week 12
  Change of SLICC/ACR score from baseline
Percentage of subjects and number of days with steroids dose equal or less to prednisone 7.5mg per day | Week 12
  Percentage of subjects and number of days with steroids dose equal or less to prednisone 7.5mg per day
Percentage of subjects with Proteinuria < 0.5g/24h in each group | Week 12
  Percentage of subjects with 24hour urine protein level less than 0.5g in each group
Percentage change of complement 3 (C3) and complement 4 (C4) from baseline in each group | Week 12
  Percentage change of complement 3 (C3) and complement 4 (C4) from baseline in each group
Percentage change of anti-dsDNA level from baseline in each group | Week 12
  Percentage change of anti-dsDNA level from baseline in each group
Time to SLE flare and Percentage of subjects with SLE flare | Baseline through week 12
  SLE flare is defined as: Compared to baseline, one new BILAG A or more than 1 new BILAG B domain score. Time to SLE flare is defined as the date of SLE flare minus the date of treatment initiation plus one.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Shen, MD & PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine affiliated Renji Hospital
Locations (1):
- Department of Rheumatology, RenJi Hospital, School of Medicine, Shanghai JiaoTong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hou LF, He SJ, Wang JX, Yang Y, Zhu FH, Zhou Y, He PL, Zhang Y, Yang YF, Li Y, Tang W, Zuo JP. SM934, a water-soluble derivative of arteminisin, exerts immunosuppressive functions in vitro and in vivo. Int Immunopharmacol. 2009 Dec;9(13-14):1509-17. doi: 10.1016/j.intimp.2009.09.003. Epub 2009 Sep 19. PMID 19772931